CLINICAL TRIAL: NCT02629250
Title: A Randomized Controlled Study of Supernormal Oxygen Delivery Goal-directed Therapy for Elderly Patients Undergoing Proximal Femoral Surgery.
Brief Title: Supernormal Oxygen Delivery for Elderly Surgical Patients
Acronym: SNODES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Xiangcai Ruan, MD, PhD, Vice-Director in Dept Anesth & Pain, Vice-Director in Dept Anesthesiology, Professor, Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GZZD-2015007
Record Dates: First submitted 2015-12-09; First posted 2015-12-14 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Femoral Fractures
Keywords: proximal femoral fracture; goal-directed therapy; myocardial injury; supernormal oxygen delivery; elders; stroke volume maximization
MeSH Terms: conditions — Femoral Fractures; Proximal Femoral Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SV maximization (Placebo Comparator): Goal-directed fluid therapy with stroke volume maximization. Device: The Volume-View system from Edwards Co.
  Interventions: Procedure: SV maximization
- supernormal DO2 (Experimental): Goal-directed fluid therapy with stroke volume maximization and supernormal oxygen delivery.
  Device: The Volume-View system from Edwards Co.
  Interventions: Procedure: supernormal DO2

INTERVENTIONS:
Procedure: SV maximization — When SpO2 ≥92%, mean arterial pressure (MAP) 65-100 mmHg, HR <100 bpm, Hb >8mg/dL and temperature ≥36℃, the patients will receive a 250 ml Ringer's lactate solution in 5 min as a fluid challenge for stroke volume (SV) maximization. The fluid challenge will repeat until the SV failed to increase by a factor of 10%. A reassessment on the SV maximization will be taken every 30 minutes and to restart algorithm when increased SV >10% or blood loss >250ml. Blood transfusions will be used to maintain a hemoglobin concentration over 8mg/dL.
  Other Names: Stroke volume maximization
  Arms: SV maximization
Procedure: supernormal DO2 — Goal directed fluid therapy is administrated as group SV maximization. Then DO2I will be assessed. If at this stage the DO2I can not be greater than 600 mL/m2 (supernormal oxygen delivery goal), then dobutamine will be started at a dose of 2.5 μg/kg/min and increased by the same increment every 20 minutes until the described target is reached or until a maximal dose of 20 μg/kg/min is given. Dobutamine is decreased in dose or discontinued if the heart rate is above 100 beats per minute or shows signs of cardiac ischemia.
  Other Names: Stroke volume maximization + supernormal oxygen delivery
  Arms: supernormal DO2

SUMMARY:
Elderly patients with poor cardiopulmonary reserve tend to suffer higher risk and develop more complications following major surgery. Quite a few researches have shown the benefits of goal-directed therapy (GDT) using fluid loading or inotropic agents or both to improve outcome during major surgery. However there is concern that inotropic therapy for a supernormal oxygen delivery (DO2I) may lead to an increased incidence of myocardial ischemia. Even though the meta-analysis has stated that DO2I strategy could possibly reduce the incidence of cardiac complication than stroke volume optimization strategy, there are very few evidence available in the literature regarding the effect on myocardial ischemia in surgical patients, especially in non-cardiac surgical patients. This study is undertaken to test the hypothesis that an intraoperative DO2I optimization result in a decreased myocardial ischemia in the elderly high-risk surgical patients.

DETAILED DESCRIPTION:
Elderly patients with poor cardiopulmonary reserve tend to suffer higher risk and develop more complications following major surgery [1]. Quite a few researches have shown the benefits of goal-directed therapy(GDT) using fluid loading or inotropic agents or both to improve outcome during major surgery [2-7]. The maintenance of adequate tissue perfusion and global oxygen delivery (DO2I) is essential to maintain adequate tissue perfusion and oxygenation in relation to increased metabolic demand during high risk surgery. However, there is concern that inotropic therapy for a supernormal oxygen delivery may lead to an increased incidence of myocardial ischemia [8]. Even though the meta-analysis has stated that DO2I optimization could possibly reduce the incidence of cardiac complication than stroke volume optimization strategy [9],there are very few evidence available in the literature regarding the effect on myocardial ischemia in surgical patients, especially in non-cardiac surgical patients. This study is undertaken to test the hypothesis that an intraoperative DO2I optimization result in a decreased myocardial ischemia in the elderly high-risk surgical patients. The investigators will conduct a prospective, randomized, controlled, double-blinded trial in seventy patients who scheduled for proximal femur surgery under General anesthesia following nerve block. Both the patients will be allocated to one of two equal groups to receive either intraoperative fluid regimen guided by SV strategy or DO2I strategy. In the control(SV) group, the patients will receive an intravenous infusion of 250 ml Ringer's lactate solution in 5 min as a fluid challenge for stroke volume maximization. In the experimental(DO2I) group, fluid and dobutamine will be given to reach a stroke volume maximization and supernormal oxygen delivery. The primary outcome is preoperative and 24h postoperative serum concentration of troponin T. Secondary outcomes include the incidence of tachycardia, arrhythmia, myocardial infarction, pneumonedema and acute heart failure, blood pressure, pulmonary infection, fluid volume, blood transfusion volume, renal function, PONV, Length of postoperative hospital stay and mortality. Data will be collected and recorded by the clinical teams who are blind to study arm allocation.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients scheduled for proximal femur fracture (PFF) surgery at this institution
2. American Society of Anaesthesiologists (ASA) physical status of III or VI
3. Two or more risk factors according to risk index of Lee

Exclusion Criteria:

1. Patient age < 70 yrs
2. Ongoing myocardial infarct or ischemia
3. Chronic haemodialysis
4. Inability to cooperate in the study
5. Patient refusal

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-02 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in concentration of troponin T at 24 hours postoperatively | preoperative value and 24 hours postoperatively
  Intraoperative supernormal oxygen delivery strategy will reduce the changes in concentration of troponin T at 24 hours postoperatively.

SECONDARY OUTCOMES:
cardiac complication up to 24 hours postoperatively | up to 24 hours postoperatively
  Occurrence of newly diagnosed arterial fibrilation ,severe arrhythmia,clinical signs of unstable angina, myocardial infarction,pulmonary edema or therapy-requiring cardiac failure.
blood pressure | up to 24 hours postoperatively
  Invasive arterial BP(mmHg) is measured through an arterial line at the arm.episode of hypotension (30% decrease in mean BP in relation to baseline values) and hypertension (30% increase in mean BP in relation to baseline values) will be recorded.
heart rate (HR) | up to 24 hours postoperatively
  HR(beats/min), bradycardia (HR < 50 beats/min), and tachycardia (HR > 100 beats/min) will be recorded at the same time as BP recording.
SpO2 | up to 24 hours postoperatively
  SpO2(%) and hypoxemia (SpO2 <90%) will be recorded at the same time as BP recording.
fluid balance | up to 24hours after surgery
  amount of fluids (ml) infused, amount of fluid losses
blood transfusion volume | up to 24 hours postoperatively
  amount of blood transfusion, amount of blood losses.
Acute Kidney Injury | up to 24 hours postoperatively
  perioperative and 24h postoperative urine volume, serum creatinine, blood urea nitrogen.
Postoperative Nausea and Vomiting (PONV) | 24 hours postoperatively
  Postoperative Nausea and Vomiting, The incidence of PONV will be recorded using a 4-point objective score (1 = no PONV;2 = mild nausea, no vomiting; 3 = excessive nausea or vomiting;4 = vomiting ≥2 times).
length of postoperative hospital stay | 28 days postoperatively
  days from end of surgery to hospital discharge
mortality | 28 days postoperatively
  mortality within 28 days after surgery
cardiac complication at 28 days postoperatively | 28 days postoperatively
  Occurrence of newly diagnosed arterial fibrilation ,severe arrhythmia,clinical signs of unstable angina, myocardial infarction,pulmonary edema or therapy-requiring cardiac failure.
incidence of pulmonary infection | up to 28 days postoperatively
  number of patients having pulmonary infection requiring intravenous antibiotic therapy

OTHER OUTCOMES:
Postoperative pain | 24 hours postoperatively
  Postoperative pain using visual analog scale (VAS, 0-100, 0 = no pain, 100 = maximum imaginable pain) will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Xiangcai Ruan, MD, PhD, Principal Investigator — Guangzhou First People's Hospital
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fowkes FG, Lunn JN, Farrow SC, Robertson IB, Samuel P. Epidemiology in anaesthesia. III: Mortality risk in patients with coexisting physical disease. Br J Anaesth. 1982 Aug;54(8):819-25. doi: 10.1093/bja/54.8.819. PMID 7104132
- [Background] Hamilton MA, Cecconi M, Rhodes A. A systematic review and meta-analysis on the use of preemptive hemodynamic intervention to improve postoperative outcomes in moderate and high-risk surgical patients. Anesth Analg. 2011 Jun;112(6):1392-402. doi: 10.1213/ANE.0b013e3181eeaae5. Epub 2010 Oct 21. PMID 20966436
- [Background] Lopes MR, Oliveira MA, Pereira VO, Lemos IP, Auler JO Jr, Michard F. Goal-directed fluid management based on pulse pressure variation monitoring during high-risk surgery: a pilot randomized controlled trial. Crit Care. 2007;11(5):R100. doi: 10.1186/cc6117. PMID 17822565
- [Background] Lobo SM, Lobo FR, Polachini CA, Patini DS, Yamamoto AE, de Oliveira NE, Serrano P, Sanches HS, Spegiorin MA, Queiroz MM, Christiano AC Jr, Savieiro EF, Alvarez PA, Teixeira SP, Cunrath GS. Prospective, randomized trial comparing fluids and dobutamine optimization of oxygen delivery in high-risk surgical patients [ISRCTN42445141]. Crit Care. 2006;10(3):R72. doi: 10.1186/cc4913. Epub 2006 May 12. PMID 16696864
- [Background] Donati A, Loggi S, Preiser JC, Orsetti G, Munch C, Gabbanelli V, Pelaia P, Pietropaoli P. Goal-directed intraoperative therapy reduces morbidity and length of hospital stay in high-risk surgical patients. Chest. 2007 Dec;132(6):1817-24. doi: 10.1378/chest.07-0621. Epub 2007 Oct 9. PMID 17925428
- [Background] Wilson J, Woods I, Fawcett J, Whall R, Dibb W, Morris C, McManus E. Reducing the risk of major elective surgery: randomised controlled trial of preoperative optimisation of oxygen delivery. BMJ. 1999 Apr 24;318(7191):1099-103. doi: 10.1136/bmj.318.7191.1099. PMID 10213716
- [Background] Pearse R, Dawson D, Fawcett J, Rhodes A, Grounds RM, Bennett ED. Early goal-directed therapy after major surgery reduces complications and duration of hospital stay. A randomised, controlled trial [ISRCTN38797445]. Crit Care. 2005;9(6):R687-93. doi: 10.1186/cc3887. Epub 2005 Nov 8. PMID 16356219
- [Background] Pearse RM, Dawson D, Fawcett J, Rhodes A, Grounds RM, Bennett D. The incidence of myocardial injury following post-operative Goal Directed Therapy. BMC Cardiovasc Disord. 2007 Mar 19;7:10. doi: 10.1186/1471-2261-7-10. PMID 17371601
- [Background] Futier E, Vallet B. Inotropes in goal-directed therapy: do we need 'goals'? Crit Care. 2010;14(5):1001. doi: 10.1186/cc9251. Epub 2010 Sep 29. PMID 20920151